CLINICAL TRIAL: NCT06675435
Title: The Effect of Inhaled Nitric Oxide on Intrapulmonary Shunt in Acutely Hypoxemic Patients With Severe Obesity
Brief Title: Inhaled Nitric Oxide in Severe Obesity
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Timothy G. Gaulton, MD, Assistant Professor of Anaesthesia, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2024p003089
Record Dates: First submitted 2024-11-04; First posted 2024-11-05 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-02

CONDITIONS: Obesity; Respiratory Insufficiency; Hypoxemic Respiratory Failure; Nitric Oxide
Keywords: severe obesity; acute hypoxemic respiratory failure; intrapulmonary shunt; inhaled nitric oxide
MeSH Terms: conditions — Obesity; Respiratory Insufficiency; Obesity, Morbid | interventions — Fractional Exhaled Nitric Oxide Testing

STUDY DESIGN:
Intervention Model Description: In a prospective single center clinical study, participants with acute hypoxemic respiratory failure will receive inhaled nitric oxide for 15 minutes. Study outcomes will compare cardiopulmonary responses to inhaled nitric oxide (vs. no inhaled nitric oxide).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Acute hypoxemic respiratory failure (Experimental): Participants (n = 40) with acute hypoxemic respiratory failure will receive inhaled nitric oxide (20 ppm) for 15 min.
  Interventions: Device: Nitric oxide
- Participants without acute hypoxemic respiratory failure (No Intervention): Participants (n = 20) without acute hypoxemic respiratory failure will not receive inhaled nitric oxide

INTERVENTIONS:
Device: Nitric oxide — 20ppm for 15 minutes delivered by INO max(Nitric Oxide) Company : INO therapeutics, Inc.
  Arms: Acute hypoxemic respiratory failure

SUMMARY:
The goal of this clinical trial is to learn about the effects of inhaled nitric oxide on oxygenation and lung perfusion in participants with severe obesity who have acute hypoxemic respiratory failure and are on mechanical ventilation

The main questions it aims to answer are:

1. In acute hypoxemic respiratory failure, what are the effects of inhaled nitric oxide on oxygenation in participants with severe obesity compared to participants with normal body weight.
2. In acute hypoxemic respiratory failure, what are the effects of inhaled nitric oxide on lung perfusion and heart function in participants with severe obesity compared to participants with normal body weight.
3. In acute hypoxemic respiratory failure, does severe obesity impact nitric oxide signaling pathways?

Participants with acute hypoxemic respiratory failure will be exposed to inhaled nitric oxide (20 ppm) while being clinically monitored.

DETAILED DESCRIPTION:
The study is a single-center, open-label clinical trial in mechanically ventilated participants with acute hypoxemic respiratory failure. The primary aim is to assess changes in intrapulmonary shunt (primary study outcome) to inhaled nitric oxide in participants with severe obesity and those with normal body weight. The secondary aims are to determine differences in regional lung perfusion (measured by electrical impedance tomography), right ventricular pressure (measured by transthoracic echocardiography), and biomarkers of nitric oxide signaling dysfunction (nitric oxide activity, pro-inflammatory cytokines, endothelial glycocalyx fragments)

The primary study intervention involves inhaled nitric oxide at 20 ppm for 15 minutes. The investigators will compare inhaled nitric oxide response in participants with severe obesity (defined by body mass index greater than or equal to 40) to participants with normal body weight (defined by body mass index 18.5-24.9). 40 participants with acute hypoxemic respiratory failure will be enrolled (20 with severe obesity and 20 with normal body weight). The investigators will enroll a separate cohort of mechanically ventilated participants who do not have acute hypoxemic respiratory failure (10 with severe obesity and 10 with normal body weight). In this cohort, investigators will collect additional blood at a single time point to compare levels of nitric oxide signaling pathways between patients with and without acute hypoxemia across body weight.

ELIGIBILITY:
For participants with acute hypoxemic respiratory failure

Inclusion Criteria:

* Acute hypoxemic respiratory failure, defined as persistent hypoxemia (PaO2/FiO2 ≤ 300 mmHg or SpO2/FiO2 ≤ 315) and on invasive mechanical ventilation for < 72 hours
* Presence of an arterial and central venous catheter (for blood gas measurement)
* Admitted to a participating MGH ICU

Exclusion Criteria:

* Age < 18 years
* Pregnancy or known active breastfeeding
* Prisoner or Incarceration
* Inability or unwillingness of subject or legal surrogate/representative to give written informed consent
* Use of inhaled or oral pulmonary vasodilatory therapy within the 24 hours preceding study enrollment
* Contraindication to inhaled NO

  * Baseline Methemoglobin ≥ 3%
  * Known left ventricle ejection fraction < 20%
  * Known history of G6PD deficiency or cytochrome issues
  * Prior adverse reaction to inhaled nitric oxide
* Presence of pneumothorax or acute pulmonary embolism
* Chronic hypoxemia requiring home supplemental non-invasive oxygen (nasal cannula or positive pressure ventilation) or home mechanical ventilation
* Chronic pulmonary vascular disease on home chemical vasodilator support (e.g., sildenafil)
* History of lung resection or transplant
* Hemodynamic instability at the time of potential study enrollment defined as:

  * Persistent systolic blood pressure < 90 mmHg or >180 mmHg despite the use of vasopressor or vasodilators or
  * Requiring an increment in inotropic-vasopressors over the past two hours just before enrollment: more than 15 mcg/min for norepinephrine and dopamine, more than 10 mcg/min in epinephrine; and more than 50 mcg/ min for phenylephrine.

EIT assessments of lung perfusion will only be performed in participants who are already receiving neuromuscular blocking agents (e.g., cisatracurium) at the time of study enrollment. EIT assessments of lung perfusion will not be performed in participants who have the following contraindications to EIT perfusion monitoring:

* Hypernatremia (serum sodium > 150 mEq/L)
* Usage of any devices with electric current generation such as pacemaker or internal cardiac defibrillator

For controls without acute hypoxemic respiratory failure

Inclusion Criteria:

* Receiving invasive mechanical ventilation and do not have a diagnosis of acute hypoxemic respiratory failure (PaO2/FiO2 > 300 mmHg or SpO2/FiO2> 315)
* Presence of an arterial catheter
* Admitted to a participating MGH ICU

Exclusion Criteria:

* Age < 18 years
* Pregnancy or known active breastfeeding
* Prisoner or Incarceration
* Inability or unwillingness of subject or legal surrogate/representative to give written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2027-10 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Intrapulmonary shunt | Intrapulmonary shunt will be assessed before inhaled nitric oxide, at 15 minutes after inhaled nitric oxide, and at 15 minutes after inhaled nitric oxide discontinuation.
  Intrapulmonary shunt will be defined as the difference in intrapulmonary shunt (%) to inhaled nitric oxide. Intrapulmonary shunt will be defined using the modified Berggren equation based on central venous and arterial oxygen concentrations from a central venous and peripheral arterial catheter.

SECONDARY OUTCOMES:
Regional pulmonary perfusion | Regional pulmonary perfusion will be assessed before inhaled nitric oxide, at 15 minutes after inhaled nitric oxide, and at 15 minutes after inhaled nitric oxide discontinuation.
  In participants who are already receiving neuromuscular blocking agents, regional pulmonary perfusion will be measured and defined as the % change to inhaled nitric oxide in 4 lung regions of interest (right upper, right lower, left upper, left lower)
Gas exchange | Gas exchange will be assessed before inhaled nitric oxide, at 15 minutes after inhaled nitric oxide, and at 15 minutes after inhaled nitric oxide discontinuation.
  Measures of gas exchange be defined by Pa02/Fi02 and dead space fraction in response to inhaled nitric oxide
Right ventricular systolic pressure | Right ventricular systolic pressure will be assessed before inhaled nitric oxide, at 15 minutes after inhaled nitric oxide, and at 15 minutes after inhaled nitric oxide discontinuation.
  The investigators will measure right ventricular systolic pressure, an ultrasound surrogate of pulmonary arterial pressure, in response to inhaled nitric oxide

OTHER OUTCOMES:
Nitric oxide activity | Nitric oxide activity will be assessed before inhaled nitric oxide, at 15 minutes after inhaled nitric oxide, and at 15 minutes after inhaled nitric oxide discontinuation. Nitric oxide activity will be measured in control participants (single timepoint).
  Nitric oxide activity will be measured by nitrate, nitrite, nitrosyl-hemoglobin using chemiluminescence in response to inhaled nitric oxide
Nitric oxide signaling pathways | Biomarkers will be measured after enrollment in participants with and without acute hypoxemic respiratory failure (single time point)
  The investigators will measure pro-inflammatory cytokines (INF-α, IL-6, IL-8, IL-10, IL-1β, TNF-α, MCP-1) using multiplex enzyme-linked immunosorbent assays and endothelial glycocalyx fragments (heparan sulfate, chondroitin sulfate, hyaluronic acid) using Liquid Chromatography (UPLC)-tandem mass spectrometry.

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Use Agreement (DUA). For more information or to submit a request, please contact the study investigators
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Data requests can be submitted starting 9 months after article publication and the data will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis.
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research.

REFERENCES:
- [Background] Spina S, Marrazzo F, Morais CCA, Victor M, Forlini C, Guarnieri M, Bastia L, Giudici R, Bassi G, Xin Y, Cereda M, Amato M, Langer T, Berra L, Fumagalli R. Modulation of pulmonary blood flow in patients with acute respiratory failure. Nitric Oxide. 2023 Jul 1;136-137:1-7. doi: 10.1016/j.niox.2023.05.001. Epub 2023 May 10. PMID 37172929
- [Background] Borges JB, Suarez-Sipmann F, Bohm SH, Tusman G, Melo A, Maripuu E, Sandstrom M, Park M, Costa EL, Hedenstierna G, Amato M. Regional lung perfusion estimated by electrical impedance tomography in a piglet model of lung collapse. J Appl Physiol (1985). 2012 Jan;112(1):225-36. doi: 10.1152/japplphysiol.01090.2010. Epub 2011 Sep 29. PMID 21960654